CLINICAL TRIAL: NCT05793671
Title: Short Term Clinical and Major Cardiovascular Adverse Events of Deferred Versus Immediate Stenting in High Thrombus Burden STEMI Patients
Brief Title: Follow up of Clinical Outcome of Deferred vs Immediate Stenting in High Thrombus Stemi Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andro thabet fawzy, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Deferred stenting in STEMI
Record Dates: First submitted 2023-03-01; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: STEMI
Keywords: STEMI patients; Heavy thrombus burden; Deferred stenting; Clinical follow up
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Closed letters will be provided in cath-lab , inside of each letter , there is a paper with decision written --> either go for stent ( for immediate stenting ) or don't go for stent ( for non-deferred stenting)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate stenting in heavy thrombus STEMI burden patients (Active Comparator): This group - heavy thrombus burden STEMI patients with thrombolysis in myocardial infarction ( TIMI ) 2-3 flow - will receive loading dose of GPIIbIIIa inhibitor intracoronary followed by immediate stenting .
  Interventions: Device: PPCI in heavy thrombus burden STEMI patients
- Deferred stenting in heavy thrombus burden STEMI patients . (Active Comparator): This group - heavy thrombus burden STEMI patients with TIMI 2-3 flow - will receive loading dose of GPIIbIIIa inhibitor intracoronary followed by GPIIbIIIa inhibitor infusion and LMWH administration for 48 -72 hours followed by stenting .
  Interventions: Device: PPCI in heavy thrombus burden STEMI patients

INTERVENTIONS:
Device: PPCI in heavy thrombus burden STEMI patients — minimally invasive procedures used to open clogged coronary arteries

SUMMARY:
To compare the effect of immediate stenting versus deferred stenting - with use of glycoproteinIIbIIIa inhibitor & low molecular weight heparin - on the clinical outcome -3 and 6 months after stenting & also infarct size using troponin level during hospital stay .

Clinical outcome - 3 and 6 months - after stenting which includes re-infarction, repeat percutaneous coronary intervention, coronary artery bypass grafting , Congestive heart failure, cardiac death & cerebrovascular accidents.

DETAILED DESCRIPTION:
Myocardial infarct¬¬¬ion is myocardial necrosis associated with impaired blood perfusion . Until now primary percutaneous coronary intervention (PPCI) is the standard modality of myocardial reperfusion However, there are a considerable number of patients whom still had acute reduction in myocardial blood perfusion after stent implantation even with patent epicardial artery which was defined as "no-reflow" That was explained by the affection of the micro-vasculature. With manipulation of culprit coronary artery lesion, distal embolization can occur, causing micro-vascular embolization & spasm which will significantly affect myocardial perfusion even with patent epicardial coronary artery Multiple methods were tried to decrease the chances of "no reflow phenomenon". Distal protection devices were used, but unfortunately with no promising results Routine thrombectomy is still controversial.

Deferred stenting, there is still controversy about the use of this strategy. At some studies, immediate stenting in thrombotic context was associated with no-reflow &distal embolization So ideas about deferred stenting started to glow when Isaac et al tried stenting deferral, after restoring culprit coronary artery patency using minimalist immediate mechanical intervention known as "MIMI - minimalist immediate mechanical intervention -" . That gave green light for further studies to explore benefits and risks of deferred stenting.

However , the strategy is still controversial , as some studies support the use of deferred stenting strategy and found it associated with better endpoints as, reduced no reflow , better myocardial perfusion and salvage lower major adverse cardiovascular events (MACE) , better left ventricular function

However there were other studies which showed no beneficial effect of deferred stenting, but even affect badly the micro-vascular obstruction. Reasons for these conflicting results included:

* Category of patients included where deferred stenting versus immediate stenting to prevent no- or slow-reflow in acute ST-segment elevation myocardial infarction (DEFER-STEMI) enrolled patients at high risk of slow flow based on clinical angiographic features, whereas DANAMI-3 DEFER was all-corner primary PCI study. A deferral strategy should only be applied after careful angiographic selection.
* DEFER-STEMI was angiographic and MRI end-point study whereas DANAMI 3-DEFER looked at clinical outcomes.
* DANAMI 3-DEFER was a larger multi-center randomized study in contrast to DEFER-STEMI.
* The use of GPIIbIIIa inhibitors in Deferred versus conventional stent implantation in patients with ST-segment elevation myocardial infarction (DANAMI 3-DEFER) was significantly lower compared to DEFERED-STEMI.
* There was high crossover to immediate stenting in the defer arm of DANAMI trial which further weakened the results.

ELIGIBILITY:
Inclusion Criteria:

* Primary percutaneous coronary intervention (PPCI) patients with culprit vessels shows heavy thrombus burden lesions.
* Culprit vessels with TIMI 2-3 either from the beginning or after MIMI (Minimalist immediate mechanical intervention).

Exclusion Criteria:

* PPCI patients with low thrombus burden lesions.
* PPCI patient with heavy thrombus burden lesions but with culprit vessels TIMI score 0-1, didn't improve after MIMI.
* patients killip II /III /IV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who develops major adverse cardiovascular events 3 months post PPCI . | 3 months post PPCI
  Major adverse cardiovascular events include re-infarction, repeat PCI, CABG, Congestive heart failure, cardiac death & CVS accidents.
Number of patients who develops major adverse cardiovascular events 6 months post PPCI . | 6 months post PPCI
  Major adverse cardiovascular events include re-infarction, repeat PCI, CABG, Congestive heart failure, cardiac death & CVS accidents.

SECONDARY OUTCOMES:
Number of patients who develop major bleeding | Within hospital admission
  major bleeding defined by bleeding in critical area , fatal bleeding , loos in hemoglobin more than 5 gm/dl .
number of patients who develop contrast induced nephropathy | Within hospital admission
  impaired renal function tests including creatinine and urea after contrast use .
Number of patients who develop allergy to tirofiban | Within hospital admission
  developing rash , angioedema , dyspnea as a reaction to tirofiban

OTHER OUTCOMES:
Number of patients who develop severe thrombocytopenia | Within hospital admission
  platelets lower than 50000 per microliter of blood

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A. Fouad, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaffe R, Charron T, Puley G, Dick A, Strauss BH. Microvascular obstruction and the no-reflow phenomenon after percutaneous coronary intervention. Circulation. 2008 Jun 17;117(24):3152-6. doi: 10.1161/CIRCULATIONAHA.107.742312. No abstract available. PMID 18559715
- [Background] Stone GW, Webb J, Cox DA, Brodie BR, Qureshi M, Kalynych A, Turco M, Schultheiss HP, Dulas D, Rutherford BD, Antoniucci D, Krucoff MW, Gibbons RJ, Jones D, Lansky AJ, Mehran R; Enhanced Myocardial Efficacy and Recovery by Aspiration of Liberated Debris (EMERALD) Investigators. Distal microcirculatory protection during percutaneous coronary intervention in acute ST-segment elevation myocardial infarction: a randomized controlled trial. JAMA. 2005 Mar 2;293(9):1063-72. doi: 10.1001/jama.293.9.1063. PMID 15741528
- [Background] Kelbaek H, Terkelsen CJ, Helqvist S, Lassen JF, Clemmensen P, Klovgaard L, Kaltoft A, Engstrom T, Botker HE, Saunamaki K, Krusell LR, Jorgensen E, Hansen HH, Christiansen EH, Ravkilde J, Kober L, Kofoed KF, Thuesen L. Randomized comparison of distal protection versus conventional treatment in primary percutaneous coronary intervention: the drug elution and distal protection in ST-elevation myocardial infarction (DEDICATION) trial. J Am Coll Cardiol. 2008 Mar 4;51(9):899-905. doi: 10.1016/j.jacc.2007.10.047. PMID 18308157
- [Background] Vlaar PJ, Svilaas T, van der Horst IC, Diercks GF, Fokkema ML, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. Lancet. 2008 Jun 7;371(9628):1915-20. doi: 10.1016/S0140-6736(08)60833-8. PMID 18539223
- [Background] Kaltoft A, Bottcher M, Nielsen SS, Hansen HH, Terkelsen C, Maeng M, Kristensen J, Thuesen L, Krusell LR, Kristensen SD, Andersen HR, Lassen JF, Rasmussen K, Rehling M, Nielsen TT, Botker HE. Routine thrombectomy in percutaneous coronary intervention for acute ST-segment-elevation myocardial infarction: a randomized, controlled trial. Circulation. 2006 Jul 4;114(1):40-7. doi: 10.1161/CIRCULATIONAHA.105.595660. Epub 2006 Jun 26. PMID 16801464
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Lim SY. No-Reflow Phoenomenon by Intracoronary Thrombus in Acute Myocardial Infarction. Chonnam Med J. 2016 Jan;52(1):38-44. doi: 10.4068/cmj.2016.52.1.38. Epub 2016 Jan 19. PMID 26865998
- [Background] Alidoosti M, Lotfi R, Lotfi-Tokaldany M, Nematipour E, Salarifar M, Poorhosseini H, Jalali A. Correlates of the "No-Reflow" or "Slow-Flow" Phenomenon in Patients Undergoing Primary Percutaneous Coronary Intervention. J Tehran Heart Cent. 2018 Jul;13(3):108-114. PMID 30745923
- [Background] Henriques JP, Zijlstra F, Ottervanger JP, de Boer MJ, van 't Hof AW, Hoorntje JC, Suryapranata H. Incidence and clinical significance of distal embolization during primary angioplasty for acute myocardial infarction. Eur Heart J. 2002 Jul;23(14):1112-7. doi: 10.1053/euhj.2001.3035. PMID 12090749
- [Background] Isaaz K, Robin C, Cerisier A, Lamaud M, Richard L, Da Costa A, Sabry MH, Gerenton C, Blanc JL. A new approach of primary angioplasty for ST-elevation acute myocardial infarction based on minimalist immediate mechanical intervention. Coron Artery Dis. 2006 May;17(3):261-9. doi: 10.1097/00019501-200605000-00010. PMID 16728877
- [Background] Ke D, Zhong W, Fan L, Chen L. Delayed versus immediate stenting for the treatment of ST-elevation acute myocardial infarction with a high thrombus burden. Coron Artery Dis. 2012 Nov;23(7):497-506. doi: 10.1097/MCA.0b013e328358a5ad. PMID 22968214
- [Background] Carrick D, Oldroyd KG, McEntegart M, Haig C, Petrie MC, Eteiba H, Hood S, Owens C, Watkins S, Layland J, Lindsay M, Peat E, Rae A, Behan M, Sood A, Hillis WS, Mordi I, Mahrous A, Ahmed N, Wilson R, Lasalle L, Genereux P, Ford I, Berry C. A randomized trial of deferred stenting versus immediate stenting to prevent no- or slow-reflow in acute ST-segment elevation myocardial infarction (DEFER-STEMI). J Am Coll Cardiol. 2014 May 27;63(20):2088-2098. doi: 10.1016/j.jacc.2014.02.530. Epub 2014 Feb 27. PMID 24583294
- [Background] Pascal J, Veugeois A, Slama M, Rahal S, Belle L, Caussin C, Amabile N. Delayed Stenting for ST-Elevation Acute Myocardial Infarction in Daily Practice: A Single-Centre Experience. Can J Cardiol. 2016 Aug;32(8):988-95. doi: 10.1016/j.cjca.2015.09.015. Epub 2015 Sep 26. PMID 26838663
- [Background] Kelbaek H, Hofsten DE, Kober L, Helqvist S, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, De Backer O, Bang LE, Kofoed KF, Lonborg J, Ahtarovski K, Vejlstrup N, Botker HE, Terkelsen CJ, Christiansen EH, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Jensen LO, Clemmensen P, Grande P, Madsen JK, Torp-Pedersen C, Engstrom T. Deferred versus conventional stent implantation in patients with ST-segment elevation myocardial infarction (DANAMI 3-DEFER): an open-label, randomised controlled trial. Lancet. 2016 May 28;387(10034):2199-206. doi: 10.1016/S0140-6736(16)30072-1. Epub 2016 Apr 3. PMID 27053444
- [Background] Belle L, Motreff P, Mangin L, Range G, Marcaggi X, Marie A, Ferrier N, Dubreuil O, Zemour G, Souteyrand G, Caussin C, Amabile N, Isaaz K, Dauphin R, Koning R, Robin C, Faurie B, Bonello L, Champin S, Delhaye C, Cuilleret F, Mewton N, Genty C, Viallon M, Bosson JL, Croisille P; MIMI Investigators*. Comparison of Immediate With Delayed Stenting Using the Minimalist Immediate Mechanical Intervention Approach in Acute ST-Segment-Elevation Myocardial Infarction: The MIMI Study. Circ Cardiovasc Interv. 2016 Mar;9(3):e003388. doi: 10.1161/CIRCINTERVENTIONS.115.003388. PMID 26957418